CLINICAL TRIAL: NCT06222749
Title: The Role of Oxytocin in Reward Processing Across the Menstrual Cycle and With Oral Contraceptive Use
Brief Title: Oxytocin and Reward Processing in Women
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: International Research Training Group 2804 (Other)
Collaborators: University Hospital Tuebingen (Other); German Research Foundation (Other); Uppsala University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Basic Science
Other Study IDs: IRTG_P06
Record Dates: First submitted 2023-12-15; First posted 2024-01-25 (Actual); Last update posted 2024-02-28 (Actual); Status verified 2024-01

CONDITIONS: Menstrual Cycle; Hormonal Contraception
Keywords: Oxytocin; Intranasal oxytocin; magnetic resonance imaging; MRI; fMRI; energy homeostasis; metabolism; reward processing; motivation; menstrual cycle; hormonal contraceptives; sex hormones; eating behavior; women's mental health
MeSH Terms: conditions — Feeding Behavior | interventions — Oxytocin

STUDY DESIGN:
Intervention Model Description: The investigators will assess the effects of oxytocin administration on reward processing and metabolism using a double-blind randomized cross-over design. In a within subject design, participants will get receive both oxytocin and placebo (both conditions) at different time points (approximately 4 weeks apart). After drug/placebo administration we will assess cerebral blood flow and functional connectivity at rest (via functional magnetic resonance imaging (fMRI)) during an effort-based decision-making task.
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: Neither participants nor investigators will know at which time point the participant will receive intranasal oxytocin and placebo. The nasal sprays will be prepared by independent members of the university hospital Tübingen.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- NC follicular (Experimental): Naturally cycling, healthy women in the follicular menstrual cycle phase.
  Interventions: Drug: Intranasal oxytocin administration; Drug: Intranasal placebo administration
- NC luteal (Experimental): Naturally cycling, healthy women in the luteal menstrual cycle phase.
  Interventions: Drug: Intranasal oxytocin administration; Drug: Intranasal placebo administration
- OC combined (Experimental): Healthy women taking combined oral hormonal contraceptives.
  Interventions: Drug: Intranasal oxytocin administration; Drug: Intranasal placebo administration
- OC progestogen-only (Experimental): Healthy women taking progestogen-only oral hormonal contraceptives.
  Interventions: Drug: Intranasal oxytocin administration; Drug: Intranasal placebo administration

INTERVENTIONS:
Drug: Intranasal oxytocin administration — 24 international units (IU) of Syntocinon, nasal spray solution; 1 ml nasal spray contains 40 I.U. oxytocin (equivalent to 67 mcg). One spray hub (0.1 ml) contains 4 I.U. oxytocin (equivalent to 6.7 mcg).
  Other Names: Syntocinon
Drug: Intranasal placebo administration — Nasal spray solution; Placebo will be administered as the placebo controlled condition.
  Other Names: Placebo

SUMMARY:
Oxytocin is a hypothalamic neuropeptide that is best known for its peripheral physiological effects in the female organism i.e., uterine contractions during birth. The neuropeptide furthermore affects reward processing and metabolic functions such as eating behavior and body weight. Oxytocin receptors are present in brain regions associated with the processing of rewards, e.g., ventral tegmental area (VTA), nucleus accumbens (NAcc) and nucleus stria terminalis.

Previous studies indicate that oxytocin interacts with sex hormones such as estradiol in a sex-specific manner. Despite known sex differences in oxytocin function, most studies i.e., on the metabolic effects of oxytocin in humans have so far focused on young, healthy men.

Intranasal oxytocin administration has emerged as a method to experimentally investigate central nervous effects of oxytocin in the absence of relevant side effects.

In the proposed study the investigators aim to systematically investigate the acute effect of intranasal oxytocin on reward processing in relation to circulating and synthetic sex hormones in healthy, naturally cycling women and in women taking hormonal oral contraceptive pills. The investigators will administer 24 international units (IU) of intranasal oxytocin vs. placebo and investigate neural correlates in a 3T MRI scanner including functional imaging during a reward processing task, changes in brain anatomy and connectivity. Additionally, metabolic functions, eating behavior and changes in mood and wellbeing will be assessed and blood will be drawn to assess parameters of hormonal and metabolic status.

DETAILED DESCRIPTION:
This pharmaco-neuroimaging study will investigate four groups of women: (1) naturally cycling (NC) women in the follicular phase of the menstrual cycle (n = 25), (2) NC women in the luteal phase of the menstrual cycle (n = 25), (3) women taking combined oral hormonal contraceptives (OC) (n = 25), (4) women taking progestogen-only OC (n = 25).

All participants will take part in an intake session (T0) and two experimental sessions (T1 and T2) scheduled approximately four weeks apart. In the intake session (T0) the eligibility of the participants i.e., MRI compatibility, will be verified. Additionally, the participants will be asked to fill out questionnaires i.e., regarding their personality, sleep and eating behavior and perform standardized cognitive tests.

To disentangle the influence of oxytocin on reward processing and metabolism across different hormonal status in females, intranasal oxytocin (24 IU) will be administered in one experimental session and placebo in another, in a randomized and double-blind study design. The investigators will obtain sex steroids (e.g., progesterone, estrogen, testosterone) i.e., to verify the menstrual cycle phase, synthetic steroids (e.g., ethinylestradiol, levonorgestrel) and metabolic hormones (e.g., glucose, insulin, c-peptide) from blood samples in the two experimental sessions. In the baseline phase of each experimental session (T1 and T2), the investigators will assess the participants body composition with bioimpedance analysis and resting energy expenditure with indirect calorimetry. After the intranasal administration of oxytocin or placebo, a 3 Tesla (3T) functional magnetic resonance imaging (fMRI) session will follow including the Effort Allocation Task (EAT), an effort-based decision-making task, a resting-state fMRI and diffusion tensor imaging (DTI) scan. The experimental sessions will furthermore assess the participants mood, thirst and hunger throughout the experimental period and include a snack test to assess eating related behavior. Additionally, participants will be asked to fill out questionnaires assessing i.e., sleep, emotion regulation, decision making, sexual function and wellbeing.

The investigators hypothesize that, (1) the acute effect of oxytocin on reward processing in naturally cycling women is most pronounced during the follicular phase and (2) the acute effect of oxytocin on reward processing in women is dampened by the intake of oral contraceptive pills (OCs), in particular progestogen-only pills.

ELIGIBILITY:
Inclusion Criteria:

* Body-mass index (BMI): 18-28 kg/m2
* Sex: female (since birth)
* Normal or corrected vision
* Natural menstrual cycle (NC) or intake of hormonal oral contraceptives (OC)
* NC: No hormonal contraception for at least 6 months; regular menstrual cycle (between 25 and 31 days) prior to participation
* OC: No hormonal contraception for at least 4 months, regular intake of OC pill

Exclusion Criteria:

* No German language fluency (due to German language test content)
* Smoking
* Medication taken within the last 6 weeks (except for OCs in the respective group)
* Current neurological or psychiatric disease (anamnestic survey)
* Current medical problems such as hormonal, metabolic, or chronic diseases (e.g., severe hypertension, diabetes, dysfunctions of the thyroid, or congestive heart failure)
* Pregnancy, delivery and lactation (current and within the last year; anamnestic survey, current pregnancy test)
* Premenstrual dysphoric disorder (PMDD), endometriosis or polycystic ovary syndrome (PCOS)
* Shift work
* NC: Any kind of hormonal treatment or contraception
* OC: Any kind of hormonal treatment or contraception (except OCs)
* Contraindication for MRI:
* Non-removable metal objects on or in the body
* Tattoos (if MRI-incompatible according to expert guidelines)
* Pathological hearing or increased sensitivity to loud noise
* Claustrophobia
* Operation less than three months ago
* Neurological disease or injury
* Moderate or severe head injury
* Intake of antidepressants or neuroleptics
* Restricted vision

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 100 (Estimated)
Dates: Start 2024-02-16 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Oxytocin and sex hormone level induced changes in reward-related brain responses in the reward circuitry during effort-based decision making. | During neuroimaging (60 minutes) oxytocin compared to placebo condition.
  Comparing brain activity (BOLD signals) in the reward circuitry (ROIs: nucleus accumbens, putamen, caudate, ventral tegmental area, amygdala, ventromedial prefrontal cortex, orbitofrontal cortex, anterior cingulate cortex, insula) and cognitive control areas (ROIs: dorsolateral and ventromedial prefrontal cortex, anterior cingulate cortex, supplementary motor area) of female participants in luteal menstrual cycle phase, follicular menstrual cycle phase, with combined OC intake and progestogen-only OC intake during a reward task with oxytocin vs placebo.
Oxytocin induced changes in reward related behavior. | During neuroimaging (60 minutes) oxytocin compared to placebo condition.
  Force exerted on grip force controller to obtain rewards and changes in behavioral parameters measured during the Effort Allocation Task after oxytocin vs. placebo administration.
Oxytocin induced changes in eating behaviour. | During the experimental session (approximately 4.5 hours).
  Number of consumed calories (kcal) in a snack test and subjective satiety in oxytocin vs. placebo condition.

SECONDARY OUTCOMES:
Oxytocin induced changes in functional connectivity. | During neuroimaging (60 minutes) oxytocin compared to placebo condition.
  Functional connectivity of regions of the mesocorticolimbic circuitry (ROIs: nucleus accumbens, putamen, caudata, ventral tegmental area, amygdala, ventral medial prefrontal cortex, orbitofrontal cortex, anterior cingulate cortex) and limbic circuity (ROIs: hypothalamus, hippocampus) after oxytocin vs. placebo administration.
Oxytocin induced changes in stress-axis reactivity. | During the experimental session (approximately 4.5 hours).
  Cortisol concentrations assessed by blood samples after oxytocin vs. placebo administration.
Sex hormone induced changes in energy expenditure. | Measured in each experimental session, approximately 4 weeks apart; between-subject outcome
  Changes in resting energy expenditure, measured by indirect calorimetry.

CONTACTS AND LOCATIONS:
Overall Officials: Manfred Hallschmid, Professor, Principal Investigator — Institute of Medical Psychology and Behavioural Neurobiology
Locations (1):
- University of Tuebingen; Department of Psychiatry & Psychotherapy; Institute of Medical Psychology and Behavioural Neurobiology, Tübingen, Baden-Wurttemberg, Germany

IPD SHARING:
Plan to Share IPD: Yes
After the publication of the key results of the study, all anonymized imaging data will be made publicly available (e.g., at openfmri.org).
Supporting Information: Study Protocol, SAP, ICF, Analytic Code
Time Frame: Data will become available after an embargo period of 12 months after completion of the study.
Access Criteria: Until the data is publicly available, researchers may contact the lead PI to gain access.